CLINICAL TRIAL: NCT02547857
Title: Transvaginal Pelvic Ultrasound in the ED
Status: Completed | Type: Observational
Sponsor: Hennepin Healthcare Research Institute (Other)
Responsible Party: Principal Investigator, Brian Driver, Associate Research Director, Hennepin Healthcare Research Institute
Other Study IDs: HSR 14-3918
Record Dates: First submitted 2015-06-15; First posted 2015-09-11 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-12

CONDITIONS: Abdominal Pain; Pelvic Pain
Keywords: Pelvic ultrasound; Transvaginal ultrasound
MeSH Terms: conditions — Abdominal Pain; Pelvic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort 1: All women who undergo pelvic US in the ED, assuming they meet inclusion/exclusion criteria
  Interventions: Other: Pelvic US

INTERVENTIONS:
Other: Pelvic US — To be eligible for inclusion, a woman will have pelvic US completed as part of her ED stay. This is a non-interventional study.

SUMMARY:
Pelvic ultrasound is frequently performed in the ED in non-pregnant women to assess for ovarian pathology, though its use has not been described in the medical literature. This observational study aims to describe its use in clinical ED practice.

DETAILED DESCRIPTION:
Pelvic ultrasound is frequently performed in the ED in non-pregnant women to assess for ovarian pathology. During the pelvic examination a transvaginal ultrasound probe is used to visualize ovarian size, determine echotexture, assess whether ovarian tenderness is present, and sometimes measure ovarian blood flow. Though pelvic ultrasound is used in the Hennepin County Medical Center ED routinely, there is a paucity of literature assessing it's utility.

This observational study will help determine the usefulness of this imaging modality, and how often it changes management in clinical practice.

Specifically, this study will attempt to determine how often transvaginal ultrasound identifies the structures of interest, and then will correlate these findings with the final ED diagnosis. If a formal ultrasound is obtained, the findings of the ED ultrasound will also be compared to the findings of the formal ultrasound.

The treating physicians will be queried the diagnosis and management plans before and after the pelvic US to ascertain changes in management.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years old female
* ED bedside transvaginal ultrasound to be performed in a non-pregnant woman with at least one ovary
* Willing to discuss how they are doing at 7-10 days via phone
* Valid phone number

Exclusion Criteria:

* If a diagnosis of ovarian torsion, mass, TOA or other ovarian pathology is known before ED ultrasound
* Previously enrolled in this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult women for whom bedside transvaginal US is planned by their treating physician will be assessed for eligibility.
Sampling Method: Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2015-09; Primary Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change in diagnosis before/after pelvic US | 8 hours (or less, this will measure what occurs during an ED stay)
  The treating physician will be queried the likelihood of EMERGENT and NON-EMERGENT ovarian pathology before and after pelvic US using the following scale: Definite, Probable, Possible, Very Unlikely. The ED tests reviewed before each of these judgements will be noted. EMERGENT is defined as ovarian torsion or tubo-ovarian abscess (TOA). NON-EMERGENT is defined as all other causes, including ovarian cyst, ovarian mass, ovarian malignancy, adnexal mass). The clinician will also free text the most likely diagnosis. A change of two or more levels (eg definite to possible, definite to very unlikely, probable to very unlikely, or vice versa) will be assumed to be a significant change in diagnosis.
Change in management plan before/after pelvic US | 8 hours (or less, this will measure what occurs during an ED stay)
  The treating physician will choose from the following regarding the management plan before/after the pelvic US: outpatient referral to OB/GYN, formal pelvic US after bedside US, consult GYN in the ED, urgent/emergent operative intervention, None of the above. Any difference in management before/after pelvic US will be considered a significant change in management.

SECONDARY OUTCOMES:
Sonographic visualization of ovaries | 8 hours (or less, this will measure what occurs during an ED stay)
  yes/no
Duration of pelvic US | 8 hours (or less, this will measure what occurs during an ED stay)
  Less than 5 minutes, 5-10 minutes, more than 10 minutes
Ovary enlargement | 8 hours (or less, this will measure what occurs during an ED stay)
  Were the ovaries larger than 3.5 x 2 cm in any plane? yes/no answer
Ovarian tenderness, sonographic | 8 hours (or less, this will measure what occurs during an ED stay)
  As a dichotomous yes/no. This will be correlated to final diagnosis. How many women with a non-tender ovary ended up with EMERGENT pathology? How many had NON-EMERGENT pathology?
Ovarian blood flow | 8 hours (or less, this will measure what occurs during an ED stay)
  The physician will determine if the ovarian flow is normal in a dichotomous yes/no answer. (if performed)
ED disposition after visit | 8 hours (or less, this will measure what occurs during an ED stay)
  This will measure if the patient is discharged from the ED or admitted to the hospital
Final ED diagnosis | 8 hours (or less, this will measure what occurs during an ED stay)
  Two questions will be answered:
  1. Ovarian Pathology, Emergency (tubo-ovarian abscess, torsion)
  2. Ovarian Pathology, Non-Emergency (cyst, mass, malignancy)
  3. Non-ovarian problem
  Question 2:
  Final ED diagnosis after all work-up: (select all that apply) checkbox
  1. ed_final_dx_2___1 ovarian cyst
  2. ed_final_dx_2___2 ovarian mass
  3. ed_final_dx_2___3 ovarian torsion
  4. ed_final_dx_2___4 tubo-ovarian abscess
  5. ed_final_dx_2___5 other ovarian pathology
  6. ed_final_dx_2___6 adnexal mass (non-ovarian)
  7. ed_final_dx_2___7 Pelvic Inflammatory Disease
  8. ed_final_dx_2___8 Abdominal pathology (appendicitis, diverticulitis, SBO, others)
  9. ed_final_dx_2___9 Non-specific abdominal pain
  10. ed_final_dx_2___10 None of the above and no ovarian pathology suspected
7-day follow-up | 7 days
  Whether another facility was visited, whether a procedure occurred, and what else happened during this stay. Patients will be attempted to be contacted three times.
Correlation between ED US and Formal US | 8 hours (or less, this will measure what occurs during an ED stay)
  If a formal US is obtained, the reading will be abstracted and compared to the ED US for the following: ovary visualization, ovary size, ovarian flow, final diagnosis, and any other abnormality in free text.
Final impression for ED ultrasound with regards to ovaries | 8 hours (or less, this will measure what occurs during an ED stay)
  NORMAL or ABNORMAL. If abnormal, the abnormality will be described.
Formal pelvic US | 8 hours (or less, this will measure what occurs during an ED stay)
  Was this study obtained? dichotomous yes/no. And why was a formal pelvic US obtained? (abnormality of ovaries on bedside US; other abnormality on bedside US; unable to visualize ovaries on bedside US; good visualization of all structures and all structures normal, but post-test probability still high; Other (free text). )The exact reason will then be listed in free text.

OTHER OUTCOMES:
Method of finding ovaries | 8 hours (or less, this will measure what occurs during an ED stay)
  Will choose from:
  1. Adjacent to pelvic vessels
  2. Followed out from uterine cornu
  3. No particular method used
Experience of sonographer | 8 hours (or less, this will measure what occurs during an ED stay)
  Choose from:
  1. G1
  2. G2
  3. G3-G5
  4. Physician Assistant (PA)
  5. Attending
  6. US tech
Pelvic physical exam characteristics | 8 hours (or less, this will measure what occurs during an ED stay)
  Was there tenderness on the exam (right/left adnexa, suprapubic region, no tenderness)? Were any masses felt? (right/left adnexa, suprapubic, no mass)

CONTACTS AND LOCATIONS:
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States